CLINICAL TRIAL: NCT06677281
Title: A Systematic Review of COVID-19's Impact on Pregnancy Outcomes
Brief Title: Impact of COVID-19 on Pregnancy Outcomes: a Systematic Review
Acronym: COVID-PREG
Status: Completed | Type: Observational
Sponsor: Zahedan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamidreza Kouhpayeh, Assistant professor, Zahedan University of Medical Sciences
Other Study IDs: COVID-PREG-2024-001
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: COVID-19; Pregnancy Outcomes; Maternal Health; Neonatal Health
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Other: Systematic Review of COVID-19's Impact on Pregnancy Outcomes — This study is a systematic review of existing literature that examines the effects of COVID-19 on pregnancy outcomes, including maternal health, neonatal health, and obstetric complications. It synthesizes data from various studies to provide an overview of the potential risks associated with COVID-19 infection during pregnancy. This intervention does not involve any new clinical trials or direct patient interaction.

SUMMARY:
This systematic review aims to evaluate the impact of COVID-19 on pregnancy outcomes. It synthesizes data from various studies to provide insights into the effects of the virus on maternal and fetal health. The review focuses on key outcomes such as preterm birth, maternal complications, and neonatal health, utilizing comprehensive literature from peer-reviewed journals. By analyzing existing studies, we aim to identify trends and gaps in research regarding COVID-19 and pregnancy. This review is intended to inform healthcare providers and pregnant individuals about potential risks and considerations during the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant individuals diagnosed with COVID-19.
* Studies reporting pregnancy outcomes related to COVID-19 published between January 2020 and the present.
* Articles that include quantitative data on maternal and fetal outcomes.

Exclusion Criteria:

* Studies that do not report on COVID-19-related pregnancy outcomes.
* Non-peer-reviewed articles or grey literature.
* Research focusing on non-pregnant populations.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of pregnant individuals diagnosed with COVID-19 as documented in various peer-reviewed studies. The review examines the impact of COVID-19 on pregnancy outcomes, including maternal health, delivery outcomes, and neonatal complications.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
Impact of COVID-19 on Maternal and Neonatal Outcomes | The review encompasses studies published from January 2020 to the present, with a focus on maternal and neonatal outcomes reported within the specified time frame.
  This primary outcome measure evaluates the various maternal and neonatal outcomes associated with COVID-19 infection during pregnancy. Key metrics include rates of maternal morbidity, neonatal morbidity, preterm birth, low birth weight, and any documented complications during pregnancy, labor, and delivery. The systematic review aims to synthesize data from available studies to provide a comprehensive understanding of these outcomes and their implications for clinical practice.

SECONDARY OUTCOMES:
Effects of COVID-19 on Pregnancy-Related Complications | The review includes data from studies published between January 2020 and the present, focusing on complications reported throughout the pregnancy and at delivery.
  This secondary outcome measure assesses the frequency and types of pregnancy-related complications associated with COVID-19. This includes conditions such as gestational hypertension, gestational diabetes, placental abruption, and other adverse effects that may arise during the pregnancy period. The review aims to analyze the incidence of these complications in pregnant individuals diagnosed with COVID-19 compared to non-infected counterparts, providing insights into how the virus may impact overall pregnancy health.

CONTACTS AND LOCATIONS:
Locations (1):
- Zahedan University of Medical Sciences, Zahedan, Sistan and Baluchestan, Iran